CLINICAL TRIAL: NCT04711005
Title: A Double-Blind, Placebo-controlled, Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and CSF Capture Study of the Safety, Pharmacokinetics and Pharmacodynamics of (2R,6R)-Hydroxynorketamine in Healthy Volunteers
Brief Title: Phase 1 Evaluation of (2R,6R)-Hydroxynorketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HNK-378227-01; 18-01 (Other: National Center for Advancing Translational Sciences (NCATS))
Record Dates: First submitted 2021-01-08; First posted 2021-01-15 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Disorder
Keywords: Healthy Volunteers; Depression; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: A 6-cohort single ascending dose (SAD) study will be conducted in healthy volunteers followed by a 2-cohort multiple ascending dose (MAD) study in healthy volunteers, followed by a 1-cohort single ascending dose study with collection of cerebrospinal fluid (CSF) and plasma for pharmacokinetics.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- SAD Cohort 1 (Experimental): (2R,6R)-Hydroxynorketamine @ 0.1 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- SAD Cohort 2 (Experimental): (2R,6R)-Hydroxynorketamine @ 0.25 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- SAD Cohort 3 (Experimental): (2R,6R)-Hydroxynorketamine @ 0.5 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- SAD Cohort 4 (Experimental): (2R,6R)-Hydroxynorketamine @ 1.0 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- SAD Cohort 5 (Experimental): (2R,6R)-Hydroxynorketamine @ 2.0 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- SAD Cohort 6 (Experimental): (2R,6R)-Hydroxynorketamine @ 4.0 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- MAD Cohort 1 (Experimental): (2R,6R)-Hydroxynorketamine @ 1.0 mg/kg via slow IV infusion (40 minutes) on days 1, 4, 7, 10
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- MAD Cohort 2 (Experimental): (2R,6R)-Hydroxynorketamine @ 2.0 mg/kg via slow IV infusion (40 minutes) on days 1, 4, 7, 10
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride
- Placebo (Placebo Comparator): Control product (placebo) will be sterile saline also administered via slow IV infusion (40 minutes).
  Interventions: Drug: Placebo
- CSF Capture Cohort 1 (Experimental): (2R,6R)-Hydroxynorketamine @ 0.25 mg/kg via slow IV infusion (40 minutes)
  Interventions: Drug: (2R,6R)-Hydroxynorketamine hydrochloride

INTERVENTIONS:
Drug: (2R,6R)-Hydroxynorketamine hydrochloride — (2R,6R)-Hydroxynorketamine is a metabolite of the drug ketamine. (2R,6R)-Hydroxynorketamine hydrochloride will be administered intravenously over a 40-minute period as a solution in a 25 mM sodium phosphate 0.9% w/v saline solution. The investigational drug product will be diluted into a 53 mL total volume of formulant.
  Arms: CSF Capture Cohort 1; MAD Cohort 1; MAD Cohort 2; SAD Cohort 1; SAD Cohort 2; SAD Cohort 3; SAD Cohort 4; SAD Cohort 5; SAD Cohort 6
Drug: Placebo — Placebo will be made up of a 0.9% w/v saline solution (53 mL total volume) administered via slow IV infusion over a 40-minute period.
  Arms: Placebo

SUMMARY:
A 6-cohort single ascending dose (SAD) study will be conducted in healthy volunteers utilizing a slow-infusion intravenous (IV) route of administration. Standard safety, pharmacokinetics (PK) and qEEG monitoring will be evaluated at all dose levels. Subsequently, a 2-cohort multiple ascending dose (MAD) study will be conducted. Doses will be administered on days 1, 4, 8, and 11. Standard safety parameters will be monitored, and PK will be evaluated at all dose levels. Finally, a single-cohort group with received a single dose by slow-infusion IV and have PK samples collected from both blood and cerebrospinal fluid (CSF).

DETAILED DESCRIPTION:
A total of 48 Subjects are planned to be enrolled in a 6-cohort SAD study (36 in the treatment groups and 12 in the control groups). All SAD cohorts will have 6 Subjects in the treatment group and 2 Subjects in placebo group. All cohorts in the SAD study will incorporate sentinel dosing which will include 1 active and 1 placebo Subject. All remaining Subjects will be dosed at least 24 hours after the sentinel cohort participants. A total of 16 Subjects are planned to be enrolled in a 2 cohort MAD study (12 in the treatment groups and 4 in the control groups). All MAD cohorts will have 6 Subjects in the treatment group and 2 Subjects in placebo group. A total of 6 subjects are planned to be enrolled in a single cohort CSF capture study. The CSF cohort will have 4 in the treatment group and 2 in the placebo group.

(2R,6R)-Hydroxynorketamine hydrochloride will be administered intravenously over a 40-minute period as a solution in a 25 mM sodium phosphate 0.9% w/v saline solution. The SAD doses will range from 0.1 mg/kg to 4.0 mg/kg and the investigational drug product will be diluted into a 53 mL total volume of formulant. Placebo will be made up of a 0.9% w/v saline solution (53 mL total volume) also administered via slow IV infusion over a 40-minute period. The MAD doses will range from 1.0 mg/kg to 2.0 mg/kg administered as a 40 minute infusion period in a solution of 25 mM sodium phosphate 0.9% w/v saline solution on days 1, 4, 8 and 11. The CSF capture doses will be 0.25 mg/mk and 2.0 mg/kg administered via slow infusion over a 40 minute period in 0.9% w/v saline solution.

Serial PK blood samples will be collected during the SAD portion for each Subject receiving drug and placebo at 9 timepoints (preinfusion, end-of-infusion [approximately 40 minutes], 1, 2, 4, 8, 12, 24, and approximately 48 hr after the start of the infusion). Pharmacokinetic urine samples will be collected during the SAD study for each Subject receiving drug and placebo at set intervals following the initiation-of-infusion (0-4, >4-8, >8-12, >12-24 hr). Serial PK blood samples will be collected for for each Subject receiving drug and placebo. Blood PK samples will be obtained at 8 timepoints for teh first and forth (last) dosing in the MAD study (preinfusion, end-of-infusion [approximately 40 minutes], 1, 2, 4, 8, 12, and approximately 24 hrs after the start of the infusion). Two PK blood samples will be collected for the second and third dosing in the MAD study for each subject receiving drug and placebo at approximately 10 minutes predose and at the end of the infusion. Serial PK blood samples will be collected for the single dose CSF capture study for each Subject receiving drug and placebo. Blood PK samples will be obtained at 8 timepoints (preinfusion, end-of-infusion [approximately 40 minutes], 1, 2, 4, 8, 12, and approximately 24hr after the start of the infusion). CSF samples will be obtained preinfusion, and at 2 timepoints (1h and 8 hours) post infusion.

Safety will be assessed throughout the study. Baseline and follow-up safety assessments will include height, body mass index (BMI), weight, temperature, medical, visual and ocular history, physical examinations, ocular examinations, visual acuity, color vision tests, electrocardiograms (ECGs), vital signs (VS), clinical laboratory tests (hematology, serum chemistry, and urinalysis), the Profile of Mood States (POMS), the Columbia-Suicide Severity Rating Scale (C-SSRS), the Clinician Administered Dissociative States Scale (CADSS), and adverse events (AEs). Safety assessments will include AEs, ECGs, VS, clinical laboratory results, and physical observations. Assessment of each Subject's level of alertness/sedation will be accomplished using the Modified Observer's Assessment of Alertness/Sedation (MOAA/S). Evaluation of safety in the MAD study will utilize the same safety assessments used in the SAD study. Evaluation of safety in the CSF capture study will utilize the same safety assessments used in the SAD and MAD study with the exception of the POMS and CADSS assessments. Monitoring of AEs will be governed by change from baselines established during prescreening and Day -1 examinations and clinical laboratory tests. Dose escalation in the SAD study or continued dosing in the MAD study may be stopped according to the predefined halting rules or if a Subject's scores demonstrate acute suicidality on the C-SSRS assessment or at the discretion of the study Principal Investigator and/or sponsor. Determination of whether to escalate to the next dose level in the SAD study or continue dosing in the MAD will be made by the Principal Investigator in consultation with the Medical Monitor and Study Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy male or female between 18 and 65 years of age (inclusive).
2. Voluntarily consents to participate in the study and provides written informed consent before the start of any study-specific procedures.
3. Be willing and able to remain in the study unit for the entire duration of the confinement period and return for outpatient visits.
4. Agree to comply with prohibitions and restrictions (section 8.5).
5. Females must have a negative serum β-human chorionic gonadotropin (hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 prior to study initiation.
6. Females must be of nonchildbearing potential or agree to use appropriate birth control, as defined in section 8.4 Contraception Requirements.
7. Males must be surgically sterile for at least 90 days before screening or agree to use a condom with spermicide when sexually active with a female partner who is not using an acceptable form of birth control during the study and for 90 days after study administration. Males must also agree to not donate sperm starting at enrollment and for 90 days after last study drug administration.
8. BMI (weight [kg]/[m2]) between 18 and 35 kg/m2 (inclusive) and weighs between 50 and 120 kg (110 - 264 pounds), inclusive.
9. Blood pressure (after Subject is in a supine position for approximately 5 minutes) between 90 and 145 mmHg systolic (inclusive) and no higher than 90 mmHg diastolic at Screening and Day -1.
10. A 12-lead ECG with no clinically significant abnormality as judged by the Investigator and QTc interval ≤ 450 milliseconds at Screening and Day -1.
11. Resting pulse rate between 45 and 100 beats per minute at Screening and Day -1.
12. Clinical laboratory findings and VS within normal range, or if outside of the normal ranges, deemed not clinically significant in the opinion of the Investigator.
13. Agree to comply with the rules regarding consumption of alcohol, caffeinated beverages, and tobacco/nicotine products during the study.

Exclusion Criteria:

1. History or presence of clinically significant medical illness including (but not limited to) hepatic, cardiovascular, pulmonary, renal, hematologic, endocrine, gastrointestinal, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease that in the opinion of the Investigator would endanger the safety of the Subject or the validity of the study results.
2. Clinically significant acute illness in the 2 weeks prior to dosing.
3. Previous or current participation in any clinical study with an investigational drug, device, or biologic within 30 days or five half-lives of the investigational product to dosing.
4. Preplanned surgery or procedures that would interfere with the conduct of the study.
5. History of severe drug or excipient allergy, or hypersensitivity to be judged at the discretion of the Investigator.
6. Donation or loss of greater than 0.5 L of blood within 90 days before screening or study start. Donation of platelets within 40 days before screening or study start. Donation of plasma within 14 days before screening or study start. Receipt of blood products within 60 days before screening or study start.
7. Recent history (2 years) of alcohol or drug abuse at the discretion of the Investigator or a positive screen for alcohol or drugs of abuse (including marijuana) at screening and upon check-in.
8. Testing positive for hepatitis B, hepatitis C, or HIV, or a history of any of these diseases. Subjects whose results are compatible with prior immunization may be included at the discretion of the Investigator.
9. History of unexplained loss of consciousness, epilepsy, or other seizure disorders, or cerebrovascular disease.
10. Malignancy within 5 years of screening visit (except basal cell or squamous cell skin carcinoma).
11. Inability to adhere to the study unit diet.
12. Use of any prescription or nonprescription medication (including vitamins, herbal preparations, and nutritional supplements) within the 14 days prior to dosing except for common analgesics (acetaminophen, ibuprofen), hormonal contraceptives or hormonal replacement therapy or nonsedating antihistamines. Topical medications may be allowed at the discretion of the Investigator.
13. History or current diagnosis of mental illness including (but not limited to) psychotic disorder, bipolar disorder, schizophrenia, borderline personality disorder, and antisocial personality disorder, generalized anxiety disorder, obsessive compulsive disorder, posttraumatic stress disorder, and eating disorders.
14. History of suicidal or homicidal ideation.
15. Significant primary sleep disorder.
16. Known allergy to ketamine, heparin, or any of the IDP components (see section 10.0 Study Drug Information).
17. Any strenuous exercise in the 2 days prior to study drug administration.
18. Consumption of beverages or food that contain alcohol, grapefruit, poppy seeds, Brussel sprouts, pomegranate, broccoli, char-grilled meat within 2 days prior to drug administration. Allowances for a single isolated incidental consumption may be evaluated and approved pending PI approval for the potential interactions.
19. Use of tobacco or nicotine-containing products within 4 weeks prior to drug administration.
20. Employee of the PI or study center with direct involvement in the proposed study or other studies under the direction of the study PI.
21. Poor peripheral venous access.
22. Close relative (parent, sibling, child) of clinical site employee.
23. Subjects who, in the opinion of the PI or designee, should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Raja, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke Early Phase Clinical Research, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2 | Placebo | CSF Capture Cohort 1
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 19 | 4
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 18 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2 | Placebo | CSF Capture Cohort 1 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 19 | 4 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 19 | 4 | 74
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (12.48) | 43.0 (16.58) | 32.5 (6.50) | 32.7 (5.01) | 29.7 (3.88) | 32.0 (6.96) | 39.0 (2.68) | 36.7 (13.28) | 37.9 (10.45) | 37.3 (13.28) | 35.4 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 4 | 1 | 2 | 3 | 3 | 7 | 2 | 30
  Male | 2 | 4 | 4 | 2 | 5 | 4 | 3 | 6 | 12 | 2 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 9
  Not Hispanic or Latino | 5 | 6 | 6 | 5 | 4 | 5 | 4 | 9 | 17 | 4 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 3 | 2 | 1 | 4 | 4 | 5 | 2 | 25
  White | 5 | 4 | 3 | 3 | 3 | 4 | 1 | 5 | 11 | 2 | 41
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 19 | 4 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability of (2R,6R)-Hydroxynorketamine
Description: Investigational product-related adverse events and serious adverse events
Time Frame: 8 days post dosing (SAD)
Population: Does not include the CSF cohorts as those were exploratory.
Measure: Count of Participants; unit: Participants
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 1 | 1 | 2

2. Primary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability of (2R,6R)-Hydroxynorketamine
Description: Investigational product-related adverse events and serious adverse events
Time Frame: 19 days post dosing (MAD)
Measure: Count of Participants; unit: Participants
Arm/Group | MAD Cohort 1 | MAD Cohort 2
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

3. Primary Outcome: Pharmacokinetics of (2R,6R)-Hydroxynorketamine, Maximum Plasma Concentration (Cmax)
Description: This parameter will be calculated as appropriate and if possible for (2R,6R)-Hydroxynorketamine, depending on actual samples collected.
Time Frame: 3 days post dosing (SAD), 11 days post dosing (MAD)
Population: Does not include the CSF cohort as that was exploratory.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 124 (31.1) | 304 (38.9) | 579 (21.3) | 1200 (26.0) | 2480 (30.3) | 4280 (16.6) | 1210 (20.8) | 2610 (13.4)

4. Primary Outcome: Pharmacokinetics of (2R,6R)-Hydroxynorketamine, Time Taken to Reach Maximum Plasma Concentration (Tmax)
Description: as for outcome 3
Time Frame: 3 days post dosing (SAD), 11 days post dosing (MAD)
Population: Does not include the CSF cohort as that was exploratory.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 0.692 [0.667 to 1.00] | 0.683 [0.617 to 1.97] | 0.692 [0.583 to 1.92] | 0.825 [0.667 to 0.983] | 0.950 [0.617 to 1.03] | 0.975 [0.617 to 1.07] | 0.667 [0.667 to 1.00] | 0.708 [0.667 to 1.00]

5. Primary Outcome: Pharmacokinetics of (2R,6R)-Hydroxynorketamine, Area Under the Curve Concentration (AUC)
Description: as for outcome 3
Time Frame: 3 days post dosing (SAD), 11 days post dosing (MAD)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 918 (22.9) | 2560 (23.5) | 5420 (15.2) | 11200 (14.5) | 19400 (15.1) | 38300 (23.7) | 9770 (10.6) | 18400 (15.1)

6. Primary Outcome: Pharmacokinetics of (2R,6R)-Hydroxynorketamine, Half-life (t1/2)
Description: as for outcome 3
Time Frame: 3 days post dosing (SAD), 11 days post dosing (MAD)
Population: Does not include the CSF cohort as that was exploratory.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 7.10 (14.9) | 7.41 (16.2) | 7.92 (8.0) | 8.18 (19.8) | 7.84 (7.9) | 6.67 (14.9) | 8.01 (14.7) | 7.60 (23)

ADVERSE EVENTS:
Time Frame: Data were collected for the SAD arms through Day 8, MAD through Day 19, CSF through Day 8, and Placebo up to Day 19.
Arm/Group | SAD Cohort 1 | SAD Cohort 2 | SAD Cohort 3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 | MAD Cohort 1 | MAD Cohort 2 | Placebo | CSF Capture Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/19 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/19 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/6 | 1/6 | 1/6 | 2/6 | 1/6 | 2/9 | 5/19 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD Cohort 1 (N=6) | SAD Cohort 2 (N=6) | SAD Cohort 3 (N=6) | SAD Cohort 4 (N=6) | SAD Cohort 5 (N=6) | SAD Cohort 6 (N=6) | MAD Cohort 1 (N=6) | MAD Cohort 2 (N=9) | Placebo (N=19) | CSF Capture Cohort 1 (N=4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diastolic blood pressure increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydratiuon (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedure site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Puncture site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in fingers (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Systolic increased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash over arms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual Disturbance (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT04711005/Prot_001.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT04711005/SAP_002.pdf
  • Informed Consent Form (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT04711005/ICF_000.pdf